CLINICAL TRIAL: NCT06359106
Title: Effects of Different Inhaled Oxygen Concentrations on Lung Function in Older Patients After Laparoscopic Gastrointestinal Surgery Under General Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wenfei Tan, Professor,Chairman, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024.3.1
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Oxygenation Index
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: 80% Oxygen (Placebo Comparator): Before anesthesia induction, the participants inhaled 100% oxygen through the mask for 3 minutes. After successful anesthesia induction, the fraction of inspired oxygen (FiO2) will be adjusted to 80%, and the total gas flow rate will be set at 2L/minute. All patients will receive treatment through the lung-protective ventilation strategy. The respiratory parameters are VT: 6-8mL/kg, positive end-expiratory pressure (PEEP), 6-8 cmH2O; RR: 1:2, and respiratory rate will be adjusted by maintaining a partial pressure of carbon dioxide at 35-45 mmHg. Manual lung recruitment maneuvers will be performed after tracheal intubation and before tracheal extubation. Blood will be collected for blood gas analysis within 48 hours after surgery.
  Interventions: Drug: 80% Oxygen
- Experimental: 40% Oxygen (Experimental): Before anesthesia induction, the participants inhaled 100% oxygen through the mask for 3 minutes. After successful anesthesia induction, FiO2 will be adjusted to 40%, and the total gas flow rate will be set at 2L/minute. All patients will receive treatment through the lung-protective ventilation strategy. The respiratory parameters are VT: 6-8mL/kg, positive end-expiratory pressure (PEEP), 6-8 cmH2O; RR: 1:2, and respiratory rate will be adjusted by maintaining a partial pressure of carbon dioxide at 35-45 mmHg. Manual lung recruitment maneuvers will be performed after tracheal intubation and before tracheal extubation. However, when intraoperative oxygen saturation is less than 94%, the manual lung recruitment maneuver will also be performed. Patients should transfer to 80% Oxygen group if intraoperative oxygen saturation less than 85%.Blood will be collected for blood gas analysis within 48 hours after surgery.
  Interventions: Drug: 40% Oxygen

INTERVENTIONS:
Drug: 80% Oxygen — After successful anesthesia induction, the fraction of inspired oxygen (FiO2) will be adjusted to 80%, and the total gas flow rate will be set at 2L/minute.
  Arms: Control: 80% Oxygen
Drug: 40% Oxygen — After successful anesthesia induction, the fraction of inspired oxygen (FiO2) will be adjusted to 40%, and the total gas flow rate will be set at 2L/minute.
  Arms: Experimental: 40% Oxygen

SUMMARY:
This was a multicenter, prospective, parallel-grouping, randomized controlled clinical study comparing low FiO2 (40%) and high FiO2 (80%) levels in older patients undergoing laparoscopic gastrointestinal surgery.

DETAILED DESCRIPTION:
This was a multicenter, prospective, parallel-grouping, randomized controlled clinical study comparing low FiO2 (40%) and high FiO2 (80%) levels in older patients undergoing laparoscopic gastrointestinal surgery. the investigators planned to enroll 1098 subjects aged > 65 years for laparoscopic gastrointestinal surgery at 19 clinical trial centers in China, randomized in a 1:1 ratio, to use two inhaled oxygen concentrations during surgery. All patients will be performed via the lung-protective ventilation strategy. The respiratory parameters are VT: 6-8ml/kg, PEEP: 6-8 cmh2O, RR: 1:2, and respiratory rate will be adjusted by maintaining a partial pressure of carbon dioxide at 35-45 mmHg. Manual lung recruitment maneuvers will be performed after tracheal intubation and before tracheal extubation. The main outcome measure was the oxygenation index on the postoperative 48h. The secondary outcome measures were the 7-day postoperative pulmonary complications and 30-day mortality rates et al.

ELIGIBILITY:
Inclusion Criteria:

* Age not less than 65 years
* American Society of Anesthesiologists grades I-III
* No history of drug allergies or abnormal anesthesia.
* The duration of mechanical ventilation was expected to be more than 2 hours.
* Laparoscopic Gastrointestinal Surgery
* The preoperative oxygen saturation was not less than 94%.
* The patients will be planned to extubate in the operating room.

Exclusion Criteria:

* History of acute lung injury or acute respiratory distress syndrome (ARDS) within 3 months.
* Cardiac function Class IV (New York Heart Association classification)
* Chronic renal failure (renal cell filtration rate <30 ml min-11.73/m2), severe liver disease
* Patients with blurred consciousness and cognitive dysfunction
* Severe coagulation dysfunction.
* Without preoperative oxygen inhalation, blood oxygen level <94%, and severe pulmonary dysfunction
* Patients with endotracheal tubes were admitted to the intensive care unit (ICU) after surgery.
* Body mass index (BMI) >30kg/m2
* Inability to complete the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1176 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Oxygenation Index | On the postoperative 48th hour
  The primary outcome was the comparison of the oxygenation index between the two groups. Oxygenation index of acute lung injury is 200, and higher scores mean worse outcome.

SECONDARY OUTCOMES:
pH value in blood gas analysis 48 hours after the operation | On the postoperative 48th hour
  pH of blood gas analysis 48 hours after the operation
oxygen inhalation time | On the postoperative 48 hour
  oxygen inhalation time
inspired oxygen concentration | On the postoperative 48 hour
  inspired oxygen concentration
oxygen uptake rate | On the postoperative 48 hour
  oxygen uptake rate
7 days pulmonary complications | On the postoperative 7th day
  7 days pulmonary complications
30-day Mortality | On the postoperative 30th day
  30-day Mortality
PaCO2 in blood gas analysis 48 hours after the operation | On the postoperative 48th hour
  PaCO2 of blood gas analysis 48 hours after the operation
Lactic acid in blood gas analysis 48 hours after the operation | On the postoperative 48th hour
  Lactic acid in blood gas analysis 48 hours after the operation

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - the First Hospital of China Medical University, Shenyang, Liaoning
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Sichuan Provincial People's Hospital, Chendu
  - Chifeng Municipal Hospital, Chifeng
  - Dalian Third People's Hospital, Dalian
  - First Affiliated Hospital, Dalian Medical University, Dalian
  - First Affiliated Hospital of Harbin Medical University, Harbin
  - Harbin Medical University Cancer Hospital, Harbin
  - First Medical University and Shandong Provincial Qianfoshan Hospital, Jinan
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Affiliated Hospital of Qingdao University, Qingdao
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Shenzhen People's Hospita, Shenzhen
  - First Hospital of Hebei Medical University, Shijia Zhuang
  - Second Hospital of Hebei Medical University, Shijia Zhuang
  - YANBIAN University Hospital（Yanbian Hospital）, Yanbian

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan will be published
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Zhang T, An Y, Zhao S, Han F, Huang L, Wang L, Wu J, Lei Q, Wang K, Shao J, Wang Y, Luan Y, Feng W, Song J, Huang Z, Wu C, Nan Y, Tang B, Sun X, Tan W. Effects of varying inhaled oxygen concentrations on lung function in older adult patients undergoing laparoscopic gastrointestinal surgery under general anesthesia: protocol of a prospective multicenter clinical study in China. Trials. 2026 Jan 23. doi: 10.1186/s13063-026-09471-3. Online ahead of print. PMID 41572351